CLINICAL TRIAL: NCT02948023
Title: Ex-vivo Cultivated Limbal Stem Cell Transplantation for Treatment of Superficial Corneal Pathologies
Brief Title: Stem Cells Therapy for Corneal Blindness
Acronym: ExCell
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: L.V. Prasad Eye Institute (Other)
Responsible Party: Principal Investigator, Vivek Singh, Dr, L.V. Prasad Eye Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LVPEI-2014-1 Version 1 15Jan14
Record Dates: First submitted 2016-10-20; First posted 2016-10-28 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Corneal Injuries; Corneal Burns; Corneal Scars and Opacities
MeSH Terms: conditions — Corneal Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Surgical therapy (No Intervention): Includes the control group that fulfills the inclusion criteria
- Ex-vivo cultivated limbal stem cell pool (Active Comparator): 0.5 million stromal and epithelial cells will be incorporated in 0.05ml of commercially available fibrin glue and pasted over the corneal lesion after epithelial debridement.
  Interventions: Biological: Ex-vivo cultivated limbal stem cell pool

INTERVENTIONS:
Biological: Ex-vivo cultivated limbal stem cell pool — 0.5 million stromal and epithelial cells will be incorporated in 0.05ml of commercially available fibrin glue and pasted over the corneal lesion after epithelial debridement.
  Arms: Ex-vivo cultivated limbal stem cell pool

SUMMARY:
This is a investigative initiated, comparative pilot clinical trial to ascertain the safety of application of ex-vivo cultivated limbal stem cells in human eyes for treating different superficial corneal pathologies. Pre-clinical work in murine models have already demonstrated efficacy of this technique in curing murine corneal pathologies.

DETAILED DESCRIPTION:
In this prospective interventional study patients with superficial corneal pathologies like scars, ulcers and burns will undergo a surgical procedure. Limbal ring from a cadaveric donor tissue, which is therapeutically accepted and serologically tested, is collected. This tissue will then be cultivated in the stem cell biology laboratory using standardized culture technique. Briefly the limbal tissue will be cut up into small pieces and digested overnight using an enzyme (Collagenase L). The cells obtained from the digest will be cultured on a petri-dish using 2% serum and growth factors. The cultured cells will be passaged three times to remove all epithelial cells from the culture. In the second procedure, the central corneal epithelium will be removed using a surgical sponge. 0.1ml of stromal cells in a concentration of 5x10^3 cells/uL diluted in the thrombin component of fibrin glue (TISEEL, Baxter) will be applied to the debrided corneal stroma. A soft bandage contact lens will be placed over the cornea at the end of the procedure. The patient will receive topical antibiotic and steroid eye drops in the post-operative period. Periodic comprehensive ophthalmic evaluation along with anterior segment optical coherence tomography (ASOCT) scanning and slit-lamp photography will be done at day 1, day 7, day 45 and day 90.

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female participants who are aged between 18-60 years.
2. Patients who are having with unilateral blindness due to superficial (defined as involving the anterior 200 microns of the corneal stroma on ASOCT imaging) corneal wounds, ulcers, burns and scars.
3. Eyes with otherwise normal.

Exclusion Criteria:

1. Active infection, proven by microbiology.
2. Unknown etiology, post-herpetic eye disease or eyes with active intra-ocular inflammation.
3. Children (<18 years of age).
4. Inability/refusal to give written informed consent or to undergo any of the anterior segment imaging tests.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-08-31 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Ocular or systemic adverse effects | until 3months after surgery

SECONDARY OUTCOMES:
Visual improvement after treatment. | until 3months after surgery
  Checking for the improvement in visual acuity that will be calculated using LogMAR chart (where 20/20 vision is normal).

CONTACTS AND LOCATIONS:
Overall Officials: Sayan Basu, MBBS, MS, Principal Investigator — LV Prasad Eye Institiute; Vivek Singh, MSc PhD, Principal Investigator — LV Prasad Eye Institiute
Locations (1):
- LV Prasad Eye Institute, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Basu S, Hertsenberg AJ, Funderburgh ML, Burrow MK, Mann MM, Du Y, Lathrop KL, Syed-Picard FN, Adams SM, Birk DE, Funderburgh JL. Human limbal biopsy-derived stromal stem cells prevent corneal scarring. Sci Transl Med. 2014 Dec 10;6(266):266ra172. doi: 10.1126/scitranslmed.3009644. PMID 25504883
- [Result] Basu S, Damala M, Singh V. Limbal Stromal Stem Cell Therapy for Acute and Chronic Superficial Corneal Pathologies: Early Clinical Outcomes of The Funderburgh Technique. Investigative Ophthalmology & Visual Science. 2017 Jun 23;58(8):3371-337

DOCUMENTS (2):
  • Study Protocol (2016-08-27): https://cdn.clinicaltrials.gov/large-docs/23/NCT02948023/Prot_000.pdf
  • Informed Consent Form (2014-01-15): https://cdn.clinicaltrials.gov/large-docs/23/NCT02948023/ICF_001.pdf